CLINICAL TRIAL: NCT03814252
Title: Prospective Clinical Safety and Efficacy Study of Lesion-targeted MRI-guided Transurethral Ultrasound Ablation for Localized Prostate Cancer
Brief Title: Prospective Clinical Safety and Efficacy Study of Lesion-targeted MRI-TULSA for Localized Prostate Cancer
Acronym: PRO-TULSA-PC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T275/2018
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Localized Prostate Cancer
Keywords: Localized prostate cancer; Transurethral ultrasound ablation; Image guided; Magnetic resonance imaging guided; Lesion-targeted; Focal therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lesion-targeted ablation with MRI-TULSA (Experimental): Intervention: Targeted lesion based thermoablation of MRI-visible biopsy proven clinically significant prostate cancer. Ablative effect is aimed to cover lesion with 5 mm MRI based healthy tissue overlap wherever possible but not compromising viability of critical tissues, mainly the wall of rectum.
  Interventions: Device: MRI-TULSA

INTERVENTIONS:
Device: MRI-TULSA — The technology is developed to ablate targeted prostate tissue through transurethrally inserted probe that transmit ultrasound energy under MRI guidance and control. The therapeutic endpoint of this method is thermal coagulation of prostate tissue.
  TULSA-PRO (Profound Medical Inc, Toronto, Canada): PAD-105, integrated into a 3 Tesla MR-system (Ingenia 3.0 Tesla, Philips Healthcare, Best, Netherlands)
  Other Names: MRI guided transurethral ultrasound ablation

SUMMARY:
Magnetic resonance imaging (MRI) has improved detection of clinically significant prostate cancer (PCa). MRI-guided transurethral ultrasound ablation (MRI-TULSA) system incorporates precise diagnosis and simultaneous ablation of prostate tissue enabling lesion-targeted treatment of PCa. Lesion-based treatment strategy spares surrounding healthy tissues from injury, which may improve the outcome of genitourinary function. This study further investigates the safety and the efficacy of lesion-targeted ablation of MRI-visible biopsy-proven PCa with MRI-TULSA.

DETAILED DESCRIPTION:
Improving diagnostic methods and screening of men with prostate specific antigen (PSA) has led to earlier detection of prostate cancer (PCa) with more favorable disease characteristics. To decrease overtreatment, low risk cases are increasingly treated with active surveillance; nevertheless some of them progress requiring interventions. Intermediate- and high-risk cases need active treatments to improve survival. However, despite desirable local control, the standard therapies including radical prostatectomy and radiation therapy, carry a risk of treatment related adverse effects to genitourinary and bowel functions. There is an eminent need for efficient PCa therapies with minimal effect on genitourinary function and quality of life. To date most studied mini-invasive technologies have used extremities of temperatures to treat PCa including high intensity focused ultrasound and cryoablation.

Magnetic resonance imaging (MRI) has improved PCa diagnosis. Novel MRI techniques enable localization and visualization of clinically significant PCa. Further, MRI can be used for guidance of targeted biopsy from suspicious lesion enhancing detection of clinically significant PCa and pinpointing a target for image guided therapies. Also, increased use of MRI may lead to more MRI-visible tumors encountered in clinical practice developing an unmet need for image guided therapies.

MRI guided transurethral ultrasound ablation (MRI-TULSA) - treatment system offers treatment strategy incorporating precise diagnosis and targeted therapy. It has been evaluated for whole-gland ablation of localized PCa. Further, lesion-targeted MRI-TULSA has been proved to be feasible and safe for treating MRI-visible-biopsy-concordant histologically significant PCa in our phase 1 treat-and-3-week-resect study (not published yet). This current study further investigates the safety and the efficacy of lesion-targeted ablation of MRI-visible biopsy-proven PCa with MRI-TULSA.

ELIGIBILITY:
Inclusion Criteria:

* Language spoken: Finnish, English or Swedish
* Mental status: Patients must be able to understand the meaning of the study
* Informed consent: The patient must sign the appropriate Ethics Committee (EC) approved informed consent documents in the presence of the designated staff.
* Biopsy-confirmed acinar adenocarcinoma of the prostate
* Gleason score ≥ 3+4/International Society of Urological Pathology grade group ≥ 2
* High volume Gleason score 6 as determined on biopsies (>2 positive cancer core or ≥ 50% cancer in a core)
* Patient presenting low volume Gleason score 6 disease and refuses active surveillance
* Non-metastatic disease; high-risk patients according to European Association of Urology risk group stratification will undergo F-Prostate specific membrane antigen-Positron Emission Tomography/Computer Tomography to exclude distant metastasis
* Lesion visible on MRI (Prostate Imaging Reporting and Data System v2 4-5)
* Eligible for general anesthesia (American Society of Anesthesiologists (ASA)≤ 3)

Exclusion Criteria:

* Contraindications for MRI (cardiac pacemaker, intracranial clips etc.)

  * Acute unresolved urinary tract infection
  * Claustrophobia
  * Hip replacement surgery or other metal in the pelvic area
  * Known allergy to gadolinium
  * Inability to insert urinary catheter
  * Suspected tumor on baseline MRI further than 30 mm or within 3 mm of the prostatic urethra
  * Prostate calcifications or cysts obstructing planned ultrasound beam path within the targeted tissue volume
  * Any other conditions that might compromise patient safety, based on the clinical judgment of the responsible urologist

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Severe adverse event free survival | 3 months
  The primary safety outcome is the freedom from severe adverse events over 3 months follow up: Clavien Dindo Classification of surgical complication is graded from 1 (mild) to 5 (death). Severe adverse events are regarded as events graded ≥3.
Oncological efficacy: Disease free survival | 12 months
  The primary oncological efficacy outcome, disease free survival (DFS), is the freedom from any histologically proven clinically significant prostate cancer as assessed from both 10-12-core systematic biopsies and MRI-directed 2-4-core in field biopsies at 12 months.

SECONDARY OUTCOMES:
Urinary continence status | 3, 6 and 12 months
  Urinary continence status as measured by Expanded Prostate Cancer Index Composite (EPIC) item 5 ≥ 2 (patient filled and reported outcome measure)
Overall urinary symptom score | 3, 6 and 12 months
  Symptom severity as measured by International Prostate Symptom Score (IPSS) (patient filled and reported outcome measure). Compared to baseline, score change of ≥ 4 is considered clinically significant.
Erectile function sufficient for penetration | 3, 6 and 12 months
  Erectile dysfunction status as measured by International Index of Erectile Function item 2 ≥ 2 (erection firmness sufficient for penetration)(patient filled and reported outcome measure). Not applicable for subject with baseline score < 2.
Overall erectile function | 3, 6 and 12 months
  Erectile function as measure by International Index of Erectile Function-5 (IIEF-5)(patient filled and reported outcome measure). Compared to baseline, score change of ≥ 4 is considered clinically significant.
Radiological failure free survival | 6 and 12 months
  Presence of a highly suspicious lesion in treatment field on prostate MRI at 6 or 12 months (Likert suspicion level ≥ 4).
Ablation failure free survival | 12 months
  In field (ablated area) biopsy-confirmed histologically viable cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Boström, M.D.Ph.D., Principal Investigator — Department of Urology, VSSHP, University of Turku
Locations (1):
- Department of Urology, VSSHP, University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fenton JJ, Weyrich MS, Durbin S, Liu Y, Bang H, Melnikow J. Prostate-Specific Antigen-Based Screening for Prostate Cancer: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2018 May 8;319(18):1914-1931. doi: 10.1001/jama.2018.3712. PMID 29801018
- [Background] Klotz L, Vesprini D, Sethukavalan P, Jethava V, Zhang L, Jain S, Yamamoto T, Mamedov A, Loblaw A. Long-term follow-up of a large active surveillance cohort of patients with prostate cancer. J Clin Oncol. 2015 Jan 20;33(3):272-7. doi: 10.1200/JCO.2014.55.1192. Epub 2014 Dec 15. PMID 25512465
- [Background] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Background] Wilt TJ, Jones KM, Barry MJ, Andriole GL, Culkin D, Wheeler T, Aronson WJ, Brawer MK. Follow-up of Prostatectomy versus Observation for Early Prostate Cancer. N Engl J Med. 2017 Jul 13;377(2):132-142. doi: 10.1056/NEJMoa1615869. PMID 28700844
- [Background] Bill-Axelson A, Holmberg L, Garmo H, Rider JR, Taari K, Busch C, Nordling S, Haggman M, Andersson SO, Spangberg A, Andren O, Palmgren J, Steineck G, Adami HO, Johansson JE. Radical prostatectomy or watchful waiting in early prostate cancer. N Engl J Med. 2014 Mar 6;370(10):932-42. doi: 10.1056/NEJMoa1311593. PMID 24597866
- [Background] Donovan JL, Hamdy FC, Lane JA, Mason M, Metcalfe C, Walsh E, Blazeby JM, Peters TJ, Holding P, Bonnington S, Lennon T, Bradshaw L, Cooper D, Herbert P, Howson J, Jones A, Lyons N, Salter E, Thompson P, Tidball S, Blaikie J, Gray C, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Davis M, Turner EL, Martin RM, Neal DE; ProtecT Study Group*. Patient-Reported Outcomes after Monitoring, Surgery, or Radiotherapy for Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1425-1437. doi: 10.1056/NEJMoa1606221. Epub 2016 Sep 14. PMID 27626365
- [Background] Valerio M, Cerantola Y, Eggener SE, Lepor H, Polascik TJ, Villers A, Emberton M. New and Established Technology in Focal Ablation of the Prostate: A Systematic Review. Eur Urol. 2017 Jan;71(1):17-34. doi: 10.1016/j.eururo.2016.08.044. Epub 2016 Aug 29. PMID 27595377
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Chin JL, Billia M, Relle J, Roethke MC, Popeneciu IV, Kuru TH, Hatiboglu G, Mueller-Wolf MB, Motsch J, Romagnoli C, Kassam Z, Harle CC, Hafron J, Nandalur KR, Chronik BA, Burtnyk M, Schlemmer HP, Pahernik S. Magnetic Resonance Imaging-Guided Transurethral Ultrasound Ablation of Prostate Tissue in Patients with Localized Prostate Cancer: A Prospective Phase 1 Clinical Trial. Eur Urol. 2016 Sep;70(3):447-55. doi: 10.1016/j.eururo.2015.12.029. Epub 2016 Jan 6. PMID 26777228
- [Background] Ramsay E, Mougenot C, Staruch R, Boyes A, Kazem M, Bronskill M, Foster H, Sugar L, Haider M, Klotz L, Chopra R. Evaluation of Focal Ablation of Magnetic Resonance Imaging Defined Prostate Cancer Using Magnetic Resonance Imaging Controlled Transurethral Ultrasound Therapy with Prostatectomy as the Reference Standard. J Urol. 2017 Jan;197(1):255-261. doi: 10.1016/j.juro.2016.06.100. Epub 2016 Aug 18. PMID 27545572
- [Background] Chopra R, Colquhoun A, Burtnyk M, N'djin WA, Kobelevskiy I, Boyes A, Siddiqui K, Foster H, Sugar L, Haider MA, Bronskill M, Klotz L. MR imaging-controlled transurethral ultrasound therapy for conformal treatment of prostate tissue: initial feasibility in humans. Radiology. 2012 Oct;265(1):303-13. doi: 10.1148/radiol.12112263. Epub 2012 Aug 28. PMID 22929332
- [Derived] Wright C, Makela P, Bigot A, Anttinen M, Bostrom PJ, Blanco Sequeiros R. Deep learning prediction of non-perfused volume without contrast agents during prostate ablation therapy. Biomed Eng Lett. 2022 Nov 8;13(1):31-40. doi: 10.1007/s13534-022-00250-y. eCollection 2023 Feb. PMID 36711157